CLINICAL TRIAL: NCT05259761
Title: Use of Unmanned Air Vehichles (Medical Drones) to Overcome Geographical Barriers to Delivery of Antiretrovial Therapy and Biological Samples.
Brief Title: Overcoming Geography With Technology: Medical Drones Project
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Makerere University (Other)
Collaborators: Johnson & Johnson (Industry); Rakai Health Sciences Program (Other)
Responsible Party: Sponsor
Other Study IDs: HREC801
Record Dates: First submitted 2021-12-14; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Sexually Transmitted Infections (Not HIV or Hepatitis); HIV Infections; COVID-19
Keywords: sample transport; anti-retroviral therapy; supply chain; unmanned ariel vehicles
MeSH Terms: conditions — Sexually Transmitted Diseases; Hepatitis; HIV Infections; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- PLHIV Kalangala District: 250 People living with HIV registered for care at Bufumira Health Centre and Mazinga Health Centre, Kalangala District
  Interventions: Other: Unmanned ariel vehicle
- NonPHLIV Kalangala District: 100 People not living with HIV attending for medical services at Bufumira Health Centre and Mazinga Health Centre, Kalangala District
  Interventions: Other: Unmanned ariel vehicle
- COVID Suspects Moyo District: 1200 people attending for COVID tests at Moyo Hospital
  Interventions: Other: Unmanned ariel vehicle

INTERVENTIONS:
Other: Unmanned ariel vehicle — Use of an Unmanned ariel vehicle for medical delivery (drugs and samples)

SUMMARY:
In this study, the investigators shall evaluate the use unmanned air vehicles (medical drones) to deliver ART to adult patients eligible/enrolled in community DSD models in Bufumira Islands, Kalangala district. The geography of the islands is ideal for this project because of the flat landscape and water coverage. The investigators hypothesize that the use of drones would be acceptable to patients and stakeholders, reduce facility drug stock outs, increase retention in care by 10% in intervention (at 12 months) compared to the control health centres and be cost neutral (to the patients and health sector perspectives). The investigators will also undertake evaluation of an efficient sample delivery system using medical drones especially for expansive rural areas like Moyo and Adjumani.

DETAILED DESCRIPTION:
Stage one will be a cross-sectional observational study with baseline data collection on ART accessibility, adherence, challenges as well as perceptions and attitudes towards possible medical drones. Stage two will be a non-randomized observational pilot of medical drones at 3 landing sites in Kalangala District, comparing to 3 landing sites without drones, and at five health facilities in Moyo and Adjumani districts. The investigators shall use qualitative and quantitative methods and a process evaluation to assess the feasibility of using drones for ART delivery and determine the impact on patient outcomes. The COVID pandemic has taken hold in Uganda since this protocol was first approved in June 2020, and having received approval from the Ministry of Health, the investigators will extend this pilot to Moyo and Adjumani Districts. The investigators shall use qualitative and quantitative methods and a process evaluation to assess the feasibility of using drones for COVID sample delivery and determine the impact on result turnaround times. Stage two includes a sub-study on validity and quality of transport of biological samples including HIV, STI, TB and COVID diagnostic and monitoring samples.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 years) or emancipated minor (15-17 years) who is HIV-infected and receiving antiretroviral therapy in Bufumira sub-county or non PLHIV adult who has attended a government health facility in Bufumira sub-county
* Resident in Kalangala district for at least the preceding 12 months with an intent to stay for a minimum next 12 months (resident is defined as those who spend more than 9 out of 12 months per year in Kalangala district, even if they move within the district)
* Evidence of a personally signed and dated informed consent document indicating that the subject (or a legal representative) has been informed of all pertinent aspects of the study.
* Willingness to comply with survey procedures

Exclusion Criteria:

* Patients with mental illness or any other medical condition that compromises decision making process.
* Any other clinical condition that, in the opinion of the site investigator, would make the participant unsuitable for the study or unable to comply with joining a DSD group.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People attending health centres in Bufumira and Mazinga sub-county will be approached for inclusion in the study. In Moyo, those with COVID symptoms will be approached.
Sampling Method: Non-Probability Sample
Enrollment: 1450 (Estimated)
Dates: Start 2021-09-22 (Actual); Primary Completion 2022-03-22 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Acceptability for ART delivery as reported using qualitative methods with key stakeholders including health care workers, district officials, people living with HIV | 24 months
  To assess acceptability of medical drone use for ART in Kalangala as compared to boat delivery through qualitative assessment including focus group discussions and in depth interviews with key stakeholders including district officials, health care workers, people living with HIV

SECONDARY OUTCOMES:
Feasibility of medical drones for ART delivery to peer support workers using number of successful flights delivering ART | 24 months
  To undertake a process evaluation for feasibility of medical drones for ART and sample transport
Retention in care as determined by attendance for ART refils at health facility or peer support group meetings in Bufumira health centre (with drone delivery) as compared to Mazinga health centre (with boat only) | 12 months
  To gather information on retention in care in PLHIV receiving ART by medical drone at 6 and 12 months in patients accessing ART compared with other ART service delivery models in Bufumira Sub County and Mazinga sub county, Kalangala District
Cost of ART transport by boat as compared to drone based on actual costs of fuel and staff time | 24 months
  To compare the cost of drone delivery compared to other ART service delivery models (e.g. individual care at health centre, outreach from health centre to landing sites, community drug distribution by boat, community drug distribution by drone) in Bufumira Sub County, Kalangala District.
Acceptability for use of medical drone to move COVID samples as reported using qualitative methods | 24 months
  To assess acceptability of medical drone use for COVID samples as compared to ground delivery through qualitative assessment including focus group discussions and in depth interviews with key stakeholders including district officials, health care workers, people who have been tested for COVID-19
Turnaround times of COVID samples from arrival in receiving laboratory to results returned to receiving laboratory delivered by medical drone as compared to by land transport | 24 months
  To compare turnaround times for samples delivered by drones as compared to delivered by land transport (standard of care) in Moyo and Adjumani districts
Cost of samples transport by medical drone as compared to by land using cost of fuel and staff time | 24 months
  To compare the cost of drone delivery compared to other sample delivery models bike or car in Moyo and Adjumani districts.

CONTACTS AND LOCATIONS:
Overall Officials: Rosalind Parkes-Ratanshi, PhD, Principal Investigator — Infectious Diseases Institute
Locations (1):
- Infectious Diseases Institute, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Informed Consent Form (2020-02-10): https://cdn.clinicaltrials.gov/large-docs/61/NCT05259761/ICF_000.pdf